CLINICAL TRIAL: NCT00206037
Title: Comparison of Open Wedge High Tibia Osteotomy Surgeries Using Colloss E and Tomofix and Tomofix Only, Regarding the Bone Healing
Brief Title: Open Wedge High Tibia Osteotomy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Interim analysis showed significant results, thus study was stopped
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Collaborators: Ossacur Inc. (Industry)
Organization: AO Innovation Translation Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-hto-colloss-05
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2007-11-20 (Estimated); Status verified 2007-11

CONDITIONS: High Tibia Osteotomy
Keywords: Tibia osteotomy; Bone healing; Bone filler; Equine Protein; COLLOSS E; TomoFix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: COLLOSS E
Device: TomoFix Plate

SUMMARY:
The aim of this RCT is to show, that in a patient group receiving COLLOSS E combined with TomoFix for medical open wedge high tibial osteotomy, the onset of bone healing is earlier in time, compared to patients receiving TomoFix without COLLOSS E.

DETAILED DESCRIPTION:
The healing effect should be demonstrated by using MRI pictures during the entire FU's in order to demonstrate the differences if COLLOSS E is applied or not.

ELIGIBILITY:
Inclusion Criteria:

* Adult and active patient
* Varus malalignment of the leg
* Intact lateral joint compartment
* Physiological age-appropriate ROM in hip, knee and ankle of affected leg

Exclusion Criteria:

* BMI>35
* Drug or alcohol abuse
* Known equine protein allergy or immunological anormalities
* Immunosuppressive treatment
* Systemic or severe local inflammation or infections
* History of active malignancy or systemic disease
* Impossible to obtain informed consent
* Legal incompetence
* Pregnant and nursing women
* Patients before, during or one year after radio- or chemotherapy
* Patients with metal or metal implants near vulnerable structures
* Patients with pacemakers or other implanted devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2005-05; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Percentage of the osteotomy gap volume filled with bone healing tissue as determined on the MRI at 2 and 6 weeks postoperatively | 6 weeks

SECONDARY OUTCOMES:
Bone union
Complication rate
Pain asset on the VAS
Deviation planing angle
Immuno reaction on equine proteins
Range of motion
Ligament stability
Time to pain free walking
WOMAC osteoarthritis index
SF36 Index

CONTACTS AND LOCATIONS:
Overall Officials: René K Marti, Prof. MD, Principal Investigator — Klinik Gut, St. Moritz
Locations (3):
- Germany (2):
  - Henriettenstiftung Hannover, Hanover
  - BGU Tuebingen, Tübingen
- Kantonsspital Luzern, Lucerne, Switzerland